CLINICAL TRIAL: NCT03425903
Title: Clinical Research, Randomized, Open, Unmasked, Controlled, Cross-group, Active-treatment, to Evaluate the Clinical Efficacy of Whole Body Cryotherapy (WBC) in the Cryosense TCT Cabin for the Treatment of Fibromyalgia
Brief Title: Evaluate the Clinical Efficacy of Whole Body Cryotherapy in the Cryosense Cabin for the Treatment of Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tecnología e Innovación Médico Estética S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TIME-CRY-2015-01
Record Dates: First submitted 2018-01-25; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia, Whole body cryotherapy
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: All participants received WBC sessions and after that become controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whole Body Cryotherapy sessions (Active Comparator): 10 Whole Body Cryotherapy sessions administered on alternate days. Patient fills the questionaires and then comes into the cabin wearing only underwear. The door is closed and the session begins, with the release of nitrogen gas to the cabin indoors, which will be in contact with the patient's body surface for 3 minutes. The intervention is performed on alternate days, so 3 sessions per week are administered. Afterwards will be compared when intervening as an control group without sessions, and with 3 visits per week and fills in the questionnaires
  Interventions: Device: Whole body cryotherapy sessions
- Control group (No Intervention): Without sessions. Patient attends a control visit weekly, for 3 consecutive weeks and fills in the questionnaires to control the variables while treatment is not applied. Afterwards will be compared when intervening as an intervention group receiving 3 sessions per week and fills in the questionnaires.

INTERVENTIONS:
Device: Whole body cryotherapy sessions — Whole body cryotherapy (WBC) 10 sessions of 3 minutes at a temperature of -196ºC (point of evaporation of liquid nitrogen), on the basis of three sessions a week.Fills in questionnaires.
  Arms: Whole Body Cryotherapy sessions

SUMMARY:
The aim of this study is to evaluate the effectiveness of an intervention with sessions of 3 minutes of whole body cryotherapy (WBC) in the Cryosense cabin. Measurement period time: 8 weeks.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effectiveness of an intervention with sessions of 3 minutes of whole body cryotherapy (WBC) in the Cryosense cabin, on the main clinical manifestations of patients with Fibromyalgia (FM).

A randomized, open and crossed 8-week clinical trial comparing a WBC intervention with the waiting list control group. Patients diagnosed with FM according to ACR 2010 criteria, in treatment and regular follow-up recruited consecutively. Two groups were made, one of intervention and one of waiting list which served as control during the first phase. At the end of the first phase, and after a week of washout, the groups crossed and went on to carry out the second phase following the opposite intervention. The pharmacological treatment was not modified during the entire study.

Trial endpoints were changed in pain after 2 and 4 weeks, measured by a visual analogue scale (VAS) and burden of disease, evaluated by the Fibromyalgia Impact Questionnaire(FIQ).

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 80 years old
* Diagnosis of Fibromyalgia according to ACR criteria
* More than 1 year from diagnosis
* Lack of response or partial response to previous treatment
* In case of women,commitment not to get pregnant during the study.

Exclusion Criteria:

* Patiens with cardiovascular or psychiatric comorbidity
* Cold intolerance
* Changes in pharmacological treatment during the study
* Body temperature over 37,5ºC

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-09 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | 8 weeks
  This instrument composed of 10 items, measures physical functioning, work status (missed days of work and job difficulty), depression, anxiety, morning tiredness, pain, stiffness, fatigue, and well-being over the past week.

SECONDARY OUTCOMES:
Combined Index of Severity of Fibromyalgia (ICAF) | 8 weeks
  Composed of 59 items, measures the combined severity index of fibromyalgia divided into 4 factors: physical, emotional, social and active and passive coping
General health questionnaire (SF36) | 8 weeks
  It´s composed of 36 questions (items) that assess both positive and negative health states
Pain intensity measure. Visual Analogyc scale (VAS) | 8 weeks
  Each patien marks in the scale the pain intensity scored 0-10 (0= no pain; 10= pain as can be)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Rivera, Doctor, Principal Investigator — Hospital Gregorio Marañón-IPR
Locations (1):
- Tecnología e Innovación Médico Estética, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rivera J, Tercero MJ, Salas JS, Gimeno JH, Alejo JS. The effect of cryotherapy on fibromyalgia: a randomised clinical trial carried out in a cryosauna cabin. Rheumatol Int. 2018 Dec;38(12):2243-2250. doi: 10.1007/s00296-018-4176-0. Epub 2018 Oct 23. PMID 30353267